CLINICAL TRIAL: NCT03849144
Title: The Effect of a Therapy Dog Activity on Employees' Stress, Mood, and Job Satisfaction and Commitment
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor and facility unable to reach agreement before study timeline expired
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Pet Partners (Unknown); Aetna, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: HM20014106
Record Dates: First submitted 2018-11-21; First posted 2019-02-21 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Stress; Mood; Job Satisfaction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapy dog activity (Experimental): Interact with visiting therapy dogs for 15 minutes on two Fridays
  Interventions: Behavioral: Therapy dog activity
- Low impact physical activity (Active Comparator): Participate in 15-minute low impact physical activity on two Fridays
  Interventions: Behavioral: Low impact exercise

INTERVENTIONS:
Behavioral: Therapy dog activity — Visiting therapy dogs and their owners, evaluated and registered as therapy dog teams with Pet Partners will be spread around a large room on the Aetna campus. Employees will arrive at scheduled times to visit with the dogs for 15 minutes, talking to the dogs and owners and petting the dogs
  Arms: Therapy dog activity
Behavioral: Low impact exercise — The low impact exercise will consist of stretching exercises conducted by a member of Aetna's wellness team in the same room for 15 minutes.
  Arms: Low impact physical activity

SUMMARY:
The goal of the current study is to determine if participating in a therapy dog activity is associated with changes in perceived stress, mood, and job satisfaction and commitment. A secondary goal is to explore a potential dose effect of multiple treatments as well as control for novelty effect.

DETAILED DESCRIPTION:
This study will be conducted at Aetna Headquarters in Hartford, Connecticut. A pre-post repeated measures design will be used to compare study participant outcomes between a treatment (therapy dog activity) and comparison (low impact physical activity) condition. Outcome variables of interest are perceived stress measured by a stress visual analog scale (SVAS), mood measured by the Positive and Negative Affect Scale (PANAS), and job satisfaction and commitment measured by an investigator-developed Job Satisfaction Survey (consisting of a combination of existing validated scales). Pet ownership, attitudes toward dogs measured by the Dog Attitude Scale, and trait stress, measured by the Perceived Stress Scale, will be assessed as moderating variables.

ELIGIBILITY:
Inclusion Criteria:

* Current Aetna employees

Exclusion Criteria:

* Individuals not employed by Aetna. Note:employees are self-selecting to participate, therefore dog fears or allergies are not listed as exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03-15 (Estimated); Primary Completion 2019-05-10 (Estimated); Study Completion 2019-07-12 (Estimated)

PRIMARY OUTCOMES:
Single Item Stress Measure | Baseline to week 3
  Changes in self reported stress on visual analog scale (VAS) immediately before and after each activity. Scale ranges from "none" to "most severe imaginable" on 15 cm scale.
20-item Positive and Negative Affect Schedule | Baseline to week 3
  Self reported mood immediately before and after each activity. Each item is scored 1-5 (1 = strongly disagree; 5 = strongly agree). 10 items comprise the positive affect scale with scores ranging from 10 - 50, with higher scores indicating higher positive affect. 10 items comprise the negative affect scale with total scores ranging from 10 - 50, with lower scores indicating lower negative affect.

SECONDARY OUTCOMES:
Single Item Stress Measure | Baseline to week 5
  Changes in self reported stress on visual analog scale (VAS) after two intervention activities. Scale ranges from "none" to "most severe imaginable" on 15 cm scale.
20-item Positive and Negative Affect Schedule | Baseline to week 5
  Self reported mood two intervention activities. Each item is scored 1-5 (1 = strongly disagree; 5 = strongly agree). 10 items comprise the positive affect scale with scores ranging from 10 - 50, with higher scores indicating higher positive affect. 10 items comprise the negative affect scale with total scores ranging from 10 - 50, with lower scores indicating lower negative affect.
9-item Job Satisfaction and Commitment Scale | Baseline to week 5
  Self reported job satisfaction ( 3 items) and commitment (6 items) at baseline, after the first and last activity. Each item is scored 1-5 (1 = strongly disagree, 5 = strongly agree). Total scores range from 9-45 with higher scores indicating greater job satisfaction and commitment

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Barker, PhD, Principal Investigator — Virginia Commonwealth University